CLINICAL TRIAL: NCT06205264
Title: Effects of Functional Strength Training at Low and High Speeds on Executive Functions in Children Aged 6-12 Years.
Brief Title: Impact of Functional Strength Training Speeds on Executive Functions in 6-12-Year-Old Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Jimenez-Roldan Manuel Jesus, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Strength_Children_EF
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Strength Training; Executive Function; Child

STUDY DESIGN:
Intervention Model Description: After the random assignment of the groups, the coaches will be oblivious to the investigation, so there is no bias.Furthermore, the principal investigator will not know where the data of each group comes from.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Group (Experimental): Effect of strength training on executive functions in children.
  Strength training sessions will have a frequency of 3 times per week (Monday, Tuesday and Wednesday) for 8 weeks. In addition, each subject is subject to an individualized training program according to the workload in order to progressively increase the intensity of work. The workload will be modified progressively by influencing both the total volume of repetitions and the intensity of the exercises. The multi joint exercises will be controlled movements and not harmful, but at maximum speed during the concentric phase of the exercise.
  Interventions: Other: Strength training at high and low speeds.
- Conventional Group (Experimental): Effect of strength training on executive functions in children.
  Strength training sessions will have a frequency of 3 times per week (Monday, Tuesday and Wednesday) for 8 weeks. In addition, each subject is subject to an individualized training program according to the workload in order to progressively increase the intensity of work. The workload will be modified progressively by influencing both the total volume of repetitions and the intensity of the exercises. This group will perform each phase of the planned exercises at a constant speed.
  Interventions: Other: Strength training at high and low speeds.

INTERVENTIONS:
Other: Strength training at high and low speeds. — The training program will last for 8 weeks with a frequency of 3 sessions per week. Session duration will be 40-60 minutes, depending on the week within the developed schedule. To form the groups, participants will be randomly divided into two groups. On one hand, the explosive group will perform exercises in less time with faster movements, while the conventional group will execute the training with slower movements. The entire session will be designed and supervised by three exercise specialists. Each child must have a written informed consent completed by their parent/guardian.
  Three days of strength training will be conducted following WHO recommendations, emphasizing multi-joint exercises.

SUMMARY:
The cognitive development in children involves fundamental changes in their thinking and understanding of the environment, enhancing skills such as attention, memory, and problem-solving. This development is linked to intelligence and mental processes, positively affecting academic performance. The prefrontal cortex, the seat of executive functions, undergoes maturation, crucial for planning and behavior regulation. Factors such as rest, language learning, and physical activity influence these functions. The study highlights the interconnection between executive functions and cognitive development in children, emphasizing the importance of early stimulation. Physical activity, especially strength training, emerges as a determinant in improving cognition and executive functions, with intensity playing a crucial role. Therefore, the aim is to investigate the effect of strength training, focusing on increased intentional execution speed compared to a constant low-speed approach.

DETAILED DESCRIPTION:
The training program will last 8 weeks and a frequency of 3 times / week.

During the week 0 the initial evaluation will be developed. Between weeks 1-8, the training program will be addressed. In week 9, all the changes made in all the measured variables will be evaluated.

Both groups will follow the same training program involving multi-joint exercises, but the Fast group will perform the concentric phase at maximum intentional speed. The Conventional Group will execute all exercises at controlled speeds.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6 and 12 years old.
* No practical contraindications for physical exercise.
* No psychological therapy.
* No mental illness.

Exclusion Criteria:

* History of Serious Musculoskeletal Injuries
* Medical Conditions Limiting Participation in Physical Activity
* Absence of Informed Consent from Parents or Guardians

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Baseline of inhibition control | Week 0
  To measure the inhibitory control, the "Stroop test" will be used. It is a short test and consists of 3 parts. In the first part they must read the greatest number of words in a sheet with a total of 100 words that appear in 5 columns. For 45 seconds they should read the largest number of words. At the end of the time the number will be written down of words read. Next, they should identify colors from a list of symbols without meaning, but colored in different colors. The subject will have to identify and name the greatest number of colors.
  Finally, the subject is given a list of words with the name of colors, but written with a different color from the one the word refers to.This test aims to assess the inhibitory control.
Mean Change from Baseline in Inhibitory control | Week 9
  To measure the inhibitory control, the "Stroop test" will be used. It is a short test and consists of 3 parts. In the first part they must read the greatest number of words in a sheet with a total of 100 words that appear in 5 columns. For 45 seconds they should read the largest number of words. At the end of the time the number will be written down of words read. Next, they should identify colors from a list of symbols without meaning, but colored in different colors. The subject will have to identify and name the greatest number of colors.
  Finally, the subject is given a list of words with the name of colors, but written with a different color from the one the word refers to.This test aims to assess the inhibitory controlof words read.

SECONDARY OUTCOMES:
Baseline of cognitive flexibility | Week 0
  To evaluate the cognitive flexibility, will be used the WISCONSIN TEST. This test consists of two sets of 64 cards. The letters present various combinations according to 4 geometric shapes, 4 colors and 4 quantities.
Mean Change from Baseline in cognitive flexibility | Week 9
  To evaluate the cognitive flexibility, will be used the WISCONSIN TEST. This test consists of two sets of 64 cards. The letters present various combinations according to 4 geometric shapes, 4 colors and 4 quantities.
Baseline of working memory | Week 0
  To evaluate working memory, the DIGIT SPAN TEST will be employed. This test involves presenting a series of numbers to the participant, who is then required to recall and repeat them in the same order (forward digit span) or in reverse order (backward digit span). The test assesses the individual's ability to temporarily store and manipulate information in their working memory. The results of the DIGIT SPAN TEST will contribute valuable insights into the impact of the strength training program on participants' cognitive functions, particularly their working memory capacity.
Mean Change from Baseline in working memory | Week 9
  To evaluate working memory, the DIGIT SPAN TEST will be employed. This test involves presenting a series of numbers to the participant, who is then required to recall and repeat them in the same order (forward digit span) or in reverse order (backward digit span). The test assesses the individual's ability to temporarily store and manipulate information in their working memory.

CONTACTS AND LOCATIONS:
Locations (1):
- Education Faculty, Seville, Spain